CLINICAL TRIAL: NCT00435019
Title: An Efficacy and Safety Comparison of Insulin Detemir vs. NPH Insulin in Children and Adolescents Diagnosed With Type 1 Diabetes
Brief Title: Comparison of NPH Insulin and Insulin Detemir in Children and Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1689; 2006-000051-18 (EudraCT Number)
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Results first posted 2009-12-08 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin detemir (Experimental): insulin detemir + insulin aspart
  Interventions: Drug: insulin detemir; Drug: insulin aspart
- NPH insulin (Experimental): NPH insulin + insulin aspart
  Interventions: Drug: insulin NPH; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin detemir — s.c. injection, once or twice daily.
  Arms: insulin detemir
Drug: insulin NPH — s.c. injection, once or twice daily.
  Arms: NPH insulin
Drug: insulin aspart — s.c. injection, at main meals.

SUMMARY:
This trial is conducted in Europe.

The aim of this research is to compare the efficacy and safety of treatment with NPH insulin and insulin detemir. You will be treated with either insulin detemir or NPH insulin once or twice daily as basal insulin. Additionally you will receive insulin aspart as bolus insulin

ELIGIBILITY:
Inclusion Criteria:

* Insulin detemir naive
* Type 1 diabetes for at least 12 months
* HbA1c lesser than or equal to 11.0%

Exclusion Criteria:

* Significant concomitant diseases

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 348 (Actual)
Dates: Start 2007-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (39):
- Bulgaria (3):
  - Novo Nordisk Investigational Site, Pleven
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Varna
- Czechia (3):
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Pardubice
  - Novo Nordisk Investigational Site, Prague
- Denmark (4):
  - Novo Nordisk Investigational Site, Glostrup Municipality
  - Novo Nordisk Investigational Site, Kolding
  - Novo Nordisk Investigational Site, Odense
  - Novo Nordisk Investigational Site, Viborg
- Finland (6):
  - Novo Nordisk Investigational Site, Espoo
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Seinäjoki
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
- France (4):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Toulouse
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Miskolc
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Poland (4):
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Kielce
  - Novo Nordisk Investigational Site, Siedlce
  - Novo Nordisk Investigational Site, Warsaw
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Turkey (Türkiye) (5):
  - Novo Nordisk Investigational Site, Altunizade-Istanbul
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir
  - Novo Nordisk Investigational Site, Kayseri
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Norfolk

REFERENCES:
- [Result] Thalange N, Bereket A, Larsen J, Hiort LC, Peterkova V. Treatment with insulin detemir or NPH insulin in children aged 2-5 yr with type 1 diabetes mellitus. Pediatr Diabetes. 2011 Nov;12(7):632-41. doi: 10.1111/j.1399-5448.2010.00750.x. Epub 2011 Mar 21. PMID 21418455
- [Result] Thalange N, Bereket A, Larsen J, Hiort LC, Peterkova V. Insulin analogues in children with Type 1 diabetes: a 52-week randomized clinical trial. Diabet Med. 2013 Feb;30(2):216-25. doi: 10.1111/dme.12041. PMID 23094597
- [Derived] Thalange N, Bereket A, Jensen LB, Hiort LC, Peterkova V. Development of Insulin Detemir/Insulin Aspart Cross-Reacting Antibodies Following Treatment with Insulin Detemir: 104-week Study in Children and Adolescents with Type 1 Diabetes Aged 2-16 Years. Diabetes Ther. 2016 Dec;7(4):713-724. doi: 10.1007/s13300-016-0196-5. Epub 2016 Sep 6. PMID 27600385
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 centres in 11 countries.
Groups:
- Insulin Detemir: Individually adjusted insulin detemir dose injected subcutaneously once daily (evening) or twice daily (morning and evening) + insulin aspart with larger meals
- NPH Insulin: Individually adjusted NPH insulin dose injected subcutaneously once daily (evening) or twice daily (morning and evening) + insulin aspart with larger meals
Period: Overall Study
Arm/Group | Insulin Detemir | NPH Insulin
Started | 177 (Randomised) | 171 (Randomised)
Exposed to Study Drug | 177 | 170 (One subject withdrew before receiving study drug, and thus not included in the full analysis set.)
Completed | 164 | 161
Not Completed | 13 | 10
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 2
Not completed — Protocol Violation | 3 | 1
Not completed — Personal reasons for withdrawal | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Detemir | NPH Insulin | Total
Number analyzed (Participants) | 177 | 170 | 347
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 177 | 170 | 347
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.0 (4.09) | 9.8 (3.90) | 9.9 (3.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 73 | 167
  Male | 83 | 97 | 180

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Haemoglobin A1c (HbA1c)
Description: Glycosylated haemoglobin A1c (HbA1c) measured after 52 weeks of treatment and analysed by central laboratory.
Time Frame: after 52 weeks of treatment
Population: Full Analysis Set (FAS) is defined as all randomised subjects exposed to at least one dose of trial product with a postbaseline observation, classified according to randomised treatment.
Measure: Mean (Standard Error); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Insulin Detemir | NPH Insulin
Number analyzed (Participants) | 171 | 168
Percent (%) glycosylated haemoglobin | 8.75 (0.11) | 8.64 (0.11)
Statistical Analysis 1: Comparison: Insulin Detemir vs NPH Insulin; Test type: Non-Inferiority or Equivalence — The null hypothesis for the non-inferiority test was that the mean HbA1c with insulin detemir was greater than or equal to the mean HbA1c with NPH insulin plus 0.4%. A sample size of 344 subjects, in total, with a drop-out rate of 20 percent would yield 274 subjects for evaluation of HbA1c. This would give 85 percent power to detect a difference in means of HbA1c of 0.4 percentage points assuming that the standard deviation was 1.1 using a two-sided t-test with a 0.05 significance level; ANCOVA; Mean Difference (Final Values) = 0.12, 95% CI [-0.12 to 0.36]

2. Secondary Outcome: Number of Subjects Reporting Adverse Events
Description: Number of subjects reporting adverse events during the trial (from week -2 to week 52).
  For details, please refer to the adverse events section.
Time Frame: from week -2 to week 52
Population: Safety analysis set (SAS): all randomised subjects exposed to at least one dose of trial product, classified according to actual treatment.
Measure: Number; unit: participants
Arm/Group | Insulin Detemir | NPH Insulin
Number analyzed (Participants) | 177 | 170
participants | 132 | 135

3. Secondary Outcome: Observed Insulin Antibody Values
Description: Observed insulin antibody values for insulin detemir specific antibodies, insulin aspart specific antibodies and insulin detemir/insulin aspart cross-reacting antibodies.
Time Frame: at 0 and 52 weeks
Population: Safety analysis set (SAS): All randomised subjects exposed to at least one dose of trial product, classified according to actual treatment. In some cases, antibody samples were taken earlier than required. These results were not included. A shipment of antibody samples was lost during transportation, and thus these antibody data were missing.
Measure: Mean (Standard Deviation); unit: Percent bound of total
Arm/Group | Insulin Detemir | NPH Insulin
Number analyzed (Participants) | 177 | 170
Percent bound of total
  Insulin detemir specific, week 0 (n=127, 112) | 3.23 (1.03) | 2.95 (1.23)
  Insulin detemir specific, week 52 (n=125, 128) | 5.15 (3.30) | 3.01 (1.66)
  Cross-reacting insulin, week 0 (n=130, 113) | 27.06 (19.1) | 27.26 (18.6)
  Cross-reacting insulin, week 52 (n=132, 135) | 43.70 (15.6) | 30.19 (17.3)
  Insulin aspart specific, week 0 (n=126, 111) | 2.26 (2.32) | 2.24 (2.99)
  Insulin aspart specific, week 52 (n=128, 133) | 4.20 (4.35) | 2.68 (3.60)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from week 0 to week 52.
Arm/Group | Insulin Detemir | NPH Insulin
Serious Adverse Events (participants affected / at risk) | 14/177 | 20/170
Other Adverse Events (participants affected / at risk) | 131/177 | 134/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=177) | NPH Insulin (N=170)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemic Unconsciousness (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Gastroenteritis (Infections and infestations) | 4 (4) | 2 (2)
Viral Infection (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis Shigella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media Acute (Infections and infestations) | 1 (1) | 0 (0)
Soft Tissue Infection (Infections and infestations) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Burns Second Degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medication Error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=177) | NPH Insulin (N=170)
Nasopharyngitis (Infections and infestations) | 75 (147) | 81 (179)
Pharyngitis (Infections and infestations) | 19 (29) | 15 (16)
Upper Respiratory Tract Infection (Infections and infestations) | 18 (32) | 16 (32)
Gastroenteritis (Infections and infestations) | 15 (20) | 12 (13)
Influenza (Infections and infestations) | 10 (14) | 18 (25)
Viral Infection (Infections and infestations) | 12 (14) | 14 (17)
Bronchitis (Infections and infestations) | 9 (11) | 12 (15)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 7 (7)
Headache (Nervous system disorders) | 26 (65) | 23 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk acknowledges the Investigator's right to publish the entire results of the trial. Any such scientific paper, presentation, communication or other information concerning the investigation described in this protocol, must be submitted in writing to Novo Nordisk Trial Manager prior to submission for publication/presentation for comments. Comments will be given within four weeks from receipt of the manuscript.